CLINICAL TRIAL: NCT00370682
Title: Phase II, Randomized, Double-blind, Single Center, Controlled Study of Two Doses of Different Formulations of the WRAIR Live Attenuated Tetravalent Dengue Vaccine Compared to a Placebo Control, Administered on a 0-6 Month Schedule, to Healthy Adults
Brief Title: A Phase II Trial of a Live Attenuated Virus Tetravalent Dengue Vaccine in Healthy Adults in Thailand
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WRAIR 1281; Study no: 103854 (T-DEN-002) (Other: GSK); HSRRB A-13699 (Other: USAMRMC)
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- T-DEN F17 (Experimental): Full Dose (0.5 mL) 0 and 6 months
  Interventions: Biological: T-DEN F17
- T-DEN F19 (Experimental): Full Dose (0.5 mL) at 0 and 6 months
  Interventions: Biological: T-DEN F-19
- Placebo Comparator (Placebo Comparator): 0.5 mL sterile buffer at 0 and 6, subcutaneous injection
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Biological: T-DEN F17 — A single dose of 0.5 mL of the dengue vaccine was injected subcutaneously into the upper-outer triceps/deltoid area of the non-dominant arm at Day 0 and at 6 months.
  Other Names: T-DEN vaccine
  Arms: T-DEN F17
Biological: T-DEN F-19 — A single dose of 0.5 mL of the dengue vaccine was injected subcutaneously into the upper-outer triceps/deltoid area of the non-dominant arm at Day 0 and at 6 months.
  Arms: T-DEN F19
Other: Placebo Comparator — A single dose of 0.5 mL of the placebo sterile solution of buffer identical in appearance to vaccine)was injected subcutaneously into the upper-outer triceps/deltoid area of the non-dominant arm at Day 0 and at 6 months.
  Arms: Placebo Comparator

SUMMARY:
This descriptive study will evaluate the safety and immunogenicity of different formulations of the WRAIR dengue vaccine compared to a placebo.

DETAILED DESCRIPTION:
Subjects will be randomized into one of three groups. One group will receive a placebo vaccine and the other two will receive different dengue vaccine formations. Each subject will receive two doses six months apart. All subjects will have 11 venipunctures during 11 visits (i.e., screening plus 10 study visits) over a period of nine months.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female adult 20-25 years of age (≥20 years of age and ≤25 years of age) at the time of vaccination;
* Free of obvious health problems as established by medical history and physical examination before entering into the study;
* Written informed consent obtained from the subject;
* Able to read the Subject Information Sheet and Consent Form;
* Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits) should be enrolled in the study;
* females must be of non-childbearing potential, i.e. surgically sterilized or, if of childbearing potential, she must be abstinent or on adequate contraceptive precautions (i.e. intrauterine contraceptive device; oral contraceptives or other equivalent hormonal contraception, e.g. progestin implantable, cutaneous hormonal patch or injectable contraceptives) for 30 days prior to vaccination, have a negative pregnancy test within 48 hours prior to vaccination and must agree to continue such precautions for 60 days after completion of the vaccination series

Exclusion Criteria:

* Pregnant or lactating female, planning to become pregnant or planning to discontinue abstinence or contraceptive precautions;
* History of any neurological or behavioral disorder or seizures, with the exception of a single febrile seizure in childhood;
* History of drug abuse or alcohol consumption (more than 2 drinks per day);
* History of allergic disease/reaction likely to be exacerbated by any component of the vaccine;
* Acute or chronic, pulmonary, cardiovascular, hepatic, renal, hematologic or endocrine functional defect, as determined by physical examination or laboratory tests;
* Any confirmed or suspected immunosuppressive or immunodeficient condition or seropositive for HBsAg, anti-HCV or anti-HIV;
* Acute disease at the time of enrollment (acute disease is defined as the presence of a moderate or severe illness with or without fever);
* Chronic hepatomegaly, right upper quadrant abdominal pain or tenderness;
* Chronic splenomegaly, left upper quadrant abdominal pain or tenderness;
* Hypertension; chest pain, palpitations, dizziness, shortness of breath, arrhythmias or friction rubs;
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the study vaccine (includes placebo) or planned use during the study period;
* Planned administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before the first dose of the study vaccine/placebo and ending 30 days after the second dose;
* A planned move to a location that will prohibit participating in the trial for 9 months after the initial vaccination;
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 90 days preceding the first dose or planned administration during the study period. For corticosteroids, this will mean prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed;
* Administration of immunoglobulins and/or blood products within 90 days preceding the first dose or planned administration during the study period;
* Any chronic systemic drug therapy to be continued during the study period (except for vitamin/mineral supplements or routine treatment for gastro-esophageal reflux);
* No easy access to a fixed or mobile telephone

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gibbons, MD, MPH, Principal Investigator — Department of Virology, Armed Forces Research Institute of Medical Sciences (AFRIMS)
Locations (1):
- Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
GSK

REFERENCES:
- [Derived] Watanaveeradej V, Gibbons RV, Simasathien S, Nisalak A, Jarman RG, Kerdpanich A, Tournay E, De La Barrerra R, Dessy F, Toussaint JF, Eckels KH, Thomas SJ, Innis BL. Safety and immunogenicity of a rederived, live-attenuated dengue virus vaccine in healthy adults living in Thailand: a randomized trial. Am J Trop Med Hyg. 2014 Jul;91(1):119-28. doi: 10.4269/ajtmh.13-0452. Epub 2014 May 27. PMID 24865677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 120 subjects were enrolled in study
Period: Overall Study
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Started | 40 | 40 | 40
Completed | 40 | 37 | 39
Not Completed | 0 | 3 | 1
Not completed — Moved from area | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.2 (1.09) | 21.7 (1.27) | 21.9 (1.19) | 21.6 (1.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 22 | 68
  Male | 17 | 17 | 18 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Southeast Asian heritage | 40 | 40 | 40 | 120
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Any Grade 3 Solicited Adverse Events (AEs) Within 21 Days Follow-up After Dose 1
Description: Percentage of subjects with any grade 3 adverse events (AEs) within 21 days follow-up after dose 1 (0 month)
Time Frame: 0-21 days after dose 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 40 | 40 | 40
percentage of subjects
  Pain | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Redness | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Swelling | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Abdominal Pain | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Arthralgia | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Fatigue | 2.5 [0.1 to 13.2] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Fever | 2.5 [0.1 to 13.2] | 0.0 [0.0 to 9.0] | 2.5 [0.1 to 13.2]
  Headache | 2.5 [0.1 to 13.2] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Mucsle Aches | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Nausea | 2.5 [0.1 to 13.2] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Pain behind eyes | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Photophobia | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Pruritus | 2.5 [0.1 to 13.2] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Rash | 5.0 [0.6 to 16.9] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]
  Vomiting | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.8]

2. Primary Outcome: Neutralizing Antibody Geometric Mean Titer (GMT) to DEN Types 1, 2, 3 and 4; 30 and 90 Days After Dose 2
Description: Neutralizing antibody geometric mean titer (GMT) to DEN types 1, 2, 3 and 4 will be measured 30 and 90 days following the administration of the 2nd dose (6 month)
Time Frame: 30 and 90 days after dose 2
Measure: Mean (95% Confidence Interval); unit: GMTs
Groups:
- PRE Dose: Pre-dose 1
- PI (M1): Post dose1 , Month 1
- PII (M7): Post dose 2, Month 7
- PII (M9): Post dose 2, Month 9
Arm/Group | PRE Dose | PI (M1) | PII (M7) | PII (M9)
Number analyzed (Participants) | 40 | 40 | 39 | 39
GMTs
  DEN-1, F17 | 172.2 [77.0 to 385.5] | 668.7 [348.1 to 1284.3] | 958.0 [606.5 to 1513.3] | 788.2 [461.9 to 1345.2]
  DEN-1, F19 | 412.6 [205.3 to 829.3] | 1111.8 [774.2 to 1596.5] | 1233.4 [914.8 to 1663.1] | 1061.1 [748.1 to 1505.1]
  DEN-1, Placebo | 412.9 [218.0 to 782.1] | 447.8 [234.5 to 855.4] | 441.8 [226.1 to 863.5] | 449.2 [240.9 to 837.6]
  DEN-2, F17 | 212.5 [99.0 to 456.2] | 860.7 [493.5 to 1501.3] | 1085.3 [803.4 to 1466.0] | 1168.7 [842.7 to 1620.9]
  DEN-2, F19 | 278.2 [132.2 to 585.6] | 1123.7 [762.9 to 1655.0] | 1274.5 [946.5 to 1716.4] | 1334.1 [1026.4 to 1734.2]
  DEN-2, Placebo | 180.3 [93.1 to 349.1] | 207.4 [106.6 to 403.3] | 216.1 [109.5 to 426.5] | 231.1 [121.1 to 441.0]
  DEN-3, F17 | 117.5 [52.7 to 261.8] | 450.2 [227.6 to 890.5] | 507.7 [288.5 to 893.6] | 519.3 [287.2 to 939.0]
  DEN-3, F19 | 241.6 [113.9 to 512.6] | 787.9 [483.5 to 1283.9] | 836.2 [514.0 to 1360.5] | 730.3 [425.1 to 1254.6]
  DEN-3, Placebo | 302.2 [154.6 to 591.0] | 289.5 [150.3 to 557.8] | 266.0 [136.5 to 518.4] | 384.7 [207.7 to 712.4]
  DEN-4, F17 | 113.7 [54.6 to 236.7] | 776.3 [470.9 to 1279.8] | 745.2 [464.5 to 1195.4] | 673.3 [419.5 to 1080.7]
  DEN-4, F19 | 149.8 [72.9 to 307.7] | 772.4 [525.1 to 1136.3] | 695.5 [467.0 to 1035.8] | 705.4 [472.8 to 1052.4]
  DEN-4, Placebo | 152.3 [80.6 to 287.5] | 158.0 [82.9 to 301.0] | 178.7 [91.7 to 348.3] | 178.4 [93.5 to 340.1]

3. Secondary Outcome: Subjects With Any Adverse Events (AEs) Within 21 Days Follow-up After Dose 2 of Study Vaccine
Description: Percentage of subjects with any adverse events (AEs) solicited and unsolicited reported during the 21-day post-vaccination period following dose 2
Time Frame: 0-21 days after dose 2 of study vaccine
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 39 | 35 | 39
percentage of subjects
  Any symptom | 74.4 [57.9 to 87.0] | 65.7 [47.8 to 80.9] | 64.1 [47.2 to 78.8]
  General symptoms | 71.8 [55.1 to 85.0] | 54.3 [36.6 to 71.2] | 53.8 [37.2 to 69.9]
  All symptoms | 51.3 [34.8 to 67.6] | 31.4 [16.9 to 49.3] | 23.1 [11.1 to 39.3]

4. Secondary Outcome: Incidence of Unsolicited AEs Within 31 Days (Days 0-30) After Any Study Vaccine Dose
Description: Incidence of unsolicited AEs reported within the 31-day (Days 0-30) post-vaccination period for each study vaccine
Time Frame: 0-30 days after each study vaccine dose
Measure: Number; unit: unsolicited AEs
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 40 | 40 | 40
unsolicited AEs | 51 | 34 | 38

5. Secondary Outcome: Incidence of Serious Adverse Events (SAEs) Throughout the Entire Study Period
Description: Number of subjects experiencing serious adverse events (SAEs) throughout the entire 9 month study period
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 40 | 40 | 40
Participants | 0 | 2 | 1

6. Secondary Outcome: Laboratory Values Above the Alert Values Within 31 Days (Days 0-30) After Each Vaccine Dose
Description: Laboratory valuesabove the alert values within 31 days (days 0-30) after each vaccine dose. Change from baseline in hematological and biochemical levels with respect to normal ranges.
  PI(D2, 5, 8, 12) = Post Dose 1, Days 2, 5, 8 and 12 PI(D5, 12,14) = Post Dose 1, Days 5, 12 and 14 PI(M1) = Post Dose 1, Month 1 PI(M6) = Post Dose 1, Month 6 PII(D2, 5, 8, 12) = Post Dose 2, Days 2, 5, 8 and 12 PII(D5, 8, 12, 14) = Post Dose 2, Days 5, 8, 12 and 14 PII(M7) = Post Dose 2, Month 7
Time Frame: within 31 days after each vaccine dose
Measure: Number; unit: subjects
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 40 | 40 | 40
subjects
  ALT - PI(D2,5,8,12) | 0 | 1 | 1
  ALT - PI(D5,12,14) | 0 | 1 | 1
  ALT - PI(M1) | 0 | 1 | 1
  AST - PI(D2,5,8,12) | 0 | 1 | 0
  AST - PI(D5,12,14) | 0 | 1 | 0
  AST - PI(M1) | 0 | 1 | 0
  AST - PI(M6) | 1 | 0 | 0
  AST - PII(D2,5,8,12) | 1 | 0 | 0
  AST - PII(D5,8,12,14) | 1 | 0 | 0
  AST - PII(M7) | 1 | 0 | 0
  Haemato-Crit - Any point | 0 | 0 | 0
  Neutro-Phil Count - PI(D2,5,8,12) | 0 | 0 | 1
  Neutro-Phil Count - PI(D5,12,14) | 0 | 0 | 1
  Neutro-Phil Count - PI(M1) | 0 | 0 | 1
  Neutro-Phil Count - PI(M6) | 0 | 1 | 1
  Neutro-Phil Count - PII(D2,5,8,12) | 0 | 1 | 1
  Neutro-Phil Count - PII(D5,8,12,14) | 0 | 1 | 1
  Neutro-Phil Count - PII(M7) | 0 | 1 | 1
  Platelets - PI(D2,5,8,12) | 0 | 1 | 2
  Platelets - PI(D5,12,14) | 0 | 1 | 2
  Platelets - PI(M1) | 0 | 1 | 2
  Platelets - PI(M6) | 0 | 0 | 2
  Platelets - PII(D2,5,8,12) | 0 | 0 | 2
  Platelets - PII(D5,8,12,14) | 0 | 0 | 2
  Platelets - PII(M7) | 0 | 0 | 2

7. Secondary Outcome: Incidence of Abnormal Findings at DEN Physical Examination After Each Vaccine Dose
Description: Incidence of abnormal dengue examination findings reported during the 31-Day (Days 0-30) post-vaccination period, per dose
Time Frame: 31 days post-vaccination per dose
Measure: Number (95% Confidence Interval); unit: % of subjects
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 40 | 40 | 40
% of subjects
  Dose 1 - Conunctival hemorrhage | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8]
  Dose 1 - Conjunctival injection | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8]
  Dose 1 - Generalized lymphadenopathy | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8]
  Dose 1 - Generalized rash | 5.0 [.06 to 16.9] | 5.0 [.06 to 16.9] | 0.0 [0.0 to 8.8]
  Dose 1 - Hepatomegaly | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8]
  Dose 1 - Lymphadenopathy | 20.0 [9.1 to 35.6] | 25.0 [12.7 to 41.2] | 25.0 [12.7 to 41.2]
  Dose 1 - Mucosal hemorrhage | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8]
  Dose 1 - Rash | 5.0 [0.6 to 16.9] | 5.0 [0.6 to 16.9] | 0.0 [0.0 to 8.8]
  Dose 1 - Skin hemorrhage | 2.5 [0.1 to 13.2] | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8]
  Dose 1 - Splenomegaly | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 8.8]
  Dose 2 - Conjunctival hemorrhage | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.3] | 0.0 [0.0 to 9.0]
  Dose 2 - Conjunctival injection | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.3] | 0.0 [0.0 to 9.0]
  Dose 2 - Generalized lymphadenopathy | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.3] | 0.0 [0.0 to 9.0]
  Dose 2 - Generalized rash | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.3] | 0.0 [0.0 to 9.0]
  Dose 2 - Hepatomegaly | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.3] | 0.0 [0.0 to 9.0]
  Dose 2 - Lymphadenopathy | 7.5 [1.6 to 20.4] | 5.3 [0.6 to 17.7] | 5.1 [0.6 to 17.3]
  Dose 2 - Mucosal hemorrhage | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.3] | 0.0 [0.0 to 9.0]
  Dose 2 - Rash | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.3] | 5.1 [0.6 to 17.3]
  Dose 2 - Skin hemorrhage | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.3] | 0.0 [0.0 to 9.0]
  Dose 2 - Splenomegaly | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 9.3] | 0.0 [0.0 to 9.0]

8. Secondary Outcome: Incidence of Suspected and Confirmed Dengue Throughout the Entire Study Period.
Description: Number of subjects with incidence of suspected and confirmed dengue throughout the entire study period.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 40 | 40 | 40
Participants | 0 | 0 | 0

9. Secondary Outcome: Percentage of Subjects With Neutralizing Antibodies to Each DEN Type, After Each Dose of Study Vaccines
Description: Percentage of subject with Tetravalent responses for neutralizing antibodies, according to pre-vaccination dengue immune status. There was no placebo run for DEN Monovalent.
  PRE = Pre-vaccination PI(M1) = Post Dose 1, Month 1 PII(M7) = Post Dose 2, Month 7
Time Frame: post dose 1 and 2
Measure: Number (95% Confidence Interval); unit: % of subjects
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 40 | 40 | 40
% of subjects
  DEN Unprimed - PRE | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18]
  DEN Unprimed - PI(M1) | 20.00 [0.51 to 71.64] | 100 [29.24 to 100] | 0.00 [0.00 to 52.18]
  DEN Unprimed - PII(M7) | 100 [47.82 to 100] | 100 [29.24 to 100] | 0.00 [0.00 to 52.18]
  DEN Monovalent - PRE | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 0.00]
  DEN Monovalent - PI(M1) | 75.00 [19.41 to 99.37] | 100 [15.81 to 100] | 0.00 [0.00 to 0.00]
  DEN Monovalent - PII(M7) | 75.00 [19.41 to 99.37] | 100 [15.81 to 100] | 0.00 [0.00 to 0.00]
  DEN Multivalent - PRE | 86.67 [69.28 to 96.24] | 90.91 [75.67 to 98.08] | 97.14 [85.08 to 99.93]
  DEN Multivalent - PI(M1) | 100 [88.43 to 100] | 100 [89.42 to 100] | 97.14 [85.08 to 99.93]
  DEN Multivalent - PII(M7) | 100 [88.43 to 100] | 100 [88.78 to 100] | 100 [89.72 to 100]

10. Secondary Outcome: Neutralizing Antibody Sero-response to Each DEN Type (Increase Neut.) Antibody From pre-to Post-vaccination, to be Determined by a Qualified Assay) After Each Dose of Study Vaccines
Description: Seropositivity rates for neut. antibodies according to pre-vaccination flavivirus immune status-primed/unprimed subjects.
  PRE = Pre-vaccination PI(M1) = Post Dose 1, Month 1 PII(M7) = Post Dose 2, Month 7 PII(M9) = Post Dose 2, Month 9
Time Frame: 9 months
Measure: Number (95% Confidence Interval); unit: % of subjects
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 40 | 40 | 40
% of subjects
  DEN-1, >10 ED50 - PRE | 76.9 [60.7 to 88.9] | 87.2 [72.6 to 95.7] | 87.5 [73.2 to 95.8]
  DEN-1, >10 ED50 - PI(M1) | 89.7 [75.8 to 97.1] | 100 [90.7 to 100] | 87.5 [73.2 to 95.8]
  DEN-1, >10 ED50 - PII(M7) | 100 [91.0 to 100] | 100 [90.3 to 100] | 87.2 [72.6 to 95.7]
  DEN-1, >10 ED50 - PII(M9) | 94.9 [82.7 to 99.4] | 100 [90.3 to 100] | 89.7 [75.8 to 97.1]
  DEN-2, >10 ED50 - PRE | 76.9 [60.7 to 88.9] | 82.1 [66.5 to 92.5] | 87.5 [73.2 to 95.8]
  DEN-2, >10 ED50 - PI(M1) | 92.3 [79.1 to 98.4] | 100 [90.7 to 100] | 87.5 [73.2 to 95.8]
  DEN-2, >10 ED50 - PII(M7) | 100 [91.0 to 100] | 100 [90.3 to 100] | 87.2 [72.6 to 95.7]
  DEN-2, >10 ED50 - PII(M9) | 100 [91.0 to 100] | 100 [90.3 to 100] | 89.7 [75.8 to 97.1]
  DEN-3, >10 ED50 - PRE | 71.8 [55.1 to 85.0] | 82.1 [66.5 to 92.5] | 85.0 [70.2 to 94.3]
  DEN-3, >10 ED50 - PI(M1) | 87.2 [72.6 to 95.7] | 100 [90.7 to 100] | 87.5 [73.2 to 95.8]
  DEN-3, >10 ED50 - PII(M7) | 97.4 [86.5 to 99.9] | 100 [90.3 to 100] | 87.2 [72.6 to 95.7]
  DEN-3, >10 ED50 - PII(M9) | 94.9 [82.7 to 99.4] | 97.2 [85.5 to 99.9] | 89.7 [75.8 to 97.1]

11. Secondary Outcome: Incidence of Measurable Dengue Viremia at Specified Time Points After Each Dose
Description: Percentage of subjects with incidence of measurable dengue viremia at specified time points after each dose.
  Negative = GEQ/uL results is equal to zero Undetermined = GEQ/uL result is below LOD Positive = GEQ/uL result is >=LOD Missing = No data PI(M1) = Post Dose 1, Month 1 PII(D2,5,8,12) = Post Dose 2, Days 2, 5,8 and 12 PII(D5,8,12,14) = Post Dose 2, Days 5, 8, 12 and 14 PII(M7) = Post Dose 2, Month 7
Time Frame: within 7 months
Measure: Number; unit: % of subjects
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
Number analyzed (Participants) | 39 | 40 | 40
% of subjects
  DEN-1, RNA - PI(D2,5,8,12): Positive | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PI(D2,5,8,12): Undetermined | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PI(D2,5,8,12): Negative | 100 | 100 | 100
  DEN-1, RNA - PI(D2,5,8,12): Missing | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PI(D5,12,14): Positive | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PI(D5,12,14): Undetermined | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PI(D5,12,14): Negative | 100 | 100 | 100
  DEN-1, RNA - PI(D5,12,14): Missing | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PI(M1): Positive | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PI(M1): Undetermined | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PI(M1): Negative | 100 | 100 | 100
  DEN-1, RNA - PI(M1): Missing | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PII(D2,5,8,12): Positive | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PII(D2,5,8,12): Undetermined | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PII(D2,5,8,12): Negative | 100 | 100 | 100
  DEN-1, RNA - PII(D2,5,8,12): Missing | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PII(D5,8,12, 14): Positive | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PII(D5,8,12, 14): Undetermined | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PII(D5,8,12, 14): Negative | 100 | 100 | 100
  DEN-1, RNA - PII(D5,8,12, 14): Missing | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PII(M7): Positive | 0.0 | 0.0 | 2.6
  DEN-1, RNA - PII(M7): Undetermined | 0.0 | 0.0 | 0.0
  DEN-1, RNA - PII(M7): Negative | 100 | 100 | 97.4
  DEN-1, RNA - PII(M7): Missing | 0.0 | 0.0 | 0.0
  DEN-2, RNA - PI(D2,5,8,12): Positive | 0.0 | 2.6 | 0.0
  DEN-2, RNA - PI(D2,5,8,12): Undetermined | 2.6 | 5.1 | 0.0
  DEN-2, RNA - PI(D2,5,8,12): Negative | 97.4 | 92.3 | 100
  DEN-2, RNA - PI(D2,5,8,12): Missing | 0.0 | 0.0 | 0.0
  DEN-2, RNA - PI(D5,12,14): Positive | 2.6 | 0.0 | 0.0
  DEN-2, RNA - PI(D5,12,14): Undetermined | 0.0 | 2.6 | 0.0
  DEN-2, RNA - PI(D5,12,14): Negative | 97.4 | 97.4 | 100
  DEN-2, RNA - PI(D5,12,14): Missing | 0.0 | 0.0 | 0.0
  DEN-2, RNA - PI(M1): Positive | 0.0 | 0.0 | 0.0
  DEN-2, RNA - PI(M1): Undetermined | 7.7 | 0.0 | 0.0
  DEN-2, RNA - PI(M1): Negative | 92.3 | 100 | 100
  DEN-2, RNA - PI(M1): Missing | 0.0 | 0.0 | 0.0
  DEN-2, RNA - PII(D2,5,8,12): Positive | 0.0 | 0.0 | 0.0
  DEN-2, RNA - PII(D2,5,8,12): Undetermined | 2.6 | 0.0 | 2.6
  DEN-2, RNA - PII(D2,5,8,12): Negative | 97.4 | 100 | 97.4
  DEN-2, RNA - PII(D2,5,8,12): Missing | 0.0 | 0.0 | 0.0
  DEN-2, RNA - PII(D5,8,12,14): Positive | 2.6 | 0.0 | 0.0
  DEN-2, RNA - PII(D5,8,12,14): Undetermined | 2.6 | 0.0 | 0.0
  DEN-2, RNA - PII(D5,8,12,14): Negative | 94.7 | 100 | 100
  DEN-2, RNA - PII(D5,8,12,14): Missing | 0.0 | 0.0 | 0.0
  DEN-2, RNA - PII(M7): Positive | 0.0 | 0.0 | 0.0
  DEN-2, RNA - PII(M7): Undetermined | 2.6 | 0.0 | 2.6
  DEN-2, RNA - PII(M7): Negative | 97.4 | 100 | 97.4
  DEN-2, RNA - PII(M7): Missing | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PI(D2,5,8,12): Positive | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PI(D2,5,8,12): Undetermined | 0.0 | 2.6 | 0.0
  DEN-3, RNA - PI(D2,5,8,12): Negative | 100 | 97.4 | 100
  DEN-3, RNA - PI(D2,5,8,12): Missing | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PI(D5,12,14): Positive | 0.0 | 2.6 | 0.0
  DEN-3, RNA - PI(D5,12,14): Undetermined | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PI(D5,12,14): Negative | 100 | 97.4 | 100
  DEN-3, RNA - PI(D5,12,14): Missing | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PI(M1): Positive | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PI(M1): Undetermined | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PI(M1): Negative | 100 | 100 | 100
  DEN-3, RNA - PI(M1): Missing | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PII(D2,5,8,12): Positive | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PII(D2,5,8,12): Undetermined | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PII(D2,5,8,12): Negative | 100 | 100 | 100
  DEN-3, RNA - PII(D2,5,8,12): Missing | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PII(D5,8,12,14): Positive | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PII(D5,8,12,14): Undetermined | 0.0 | 0.0 | 2.6
  DEN-3, RNA - PII(D5,8,12,14): Negative | 100 | 100 | 97.4
  DEN-3, RNA - PII(D5,8,12,14): Missing | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PII(M7): Positive | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PII(M7): Undetermined | 0.0 | 0.0 | 0.0
  DEN-3, RNA - PII(M7): Negative | 100 | 100 | 100
  DEN-3, RNA - PII(M7): Missing | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PI(D2,5,8,12): Positive | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PI(D2,5,8,12): Undetermined | 2.6 | 0.0 | 0.0
  DEN-4, RNA - PI(D2,5,8,12): Negative | 97.4 | 100 | 100
  DEN-4, RNA - PI(D2,5,8,12): Missing | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PI(D5,12,14): Positive | 2.6 | 0.0 | 0.0
  DEN-4, RNA - PI(D5,12,14): Undetermined | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PI(D5,12,14): Negative | 97.4 | 100 | 100
  DEN-4, RNA - PI(D5,12,14): Missing | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PI(M1): Positive | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PI(M1): Undetermined | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PI(M1): Negative | 100 | 100 | 100
  DEN-4, RNA - PI(M1): Missing | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PII(D2,5,8,12): Positive | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PII(D2,5,8,12): Undetermined | 0.0 | 2.9 | 0.0
  DEN-4, RNA - PII(D2,5,8,12): Negative | 100 | 97.1 | 100
  DEN-4, RNA - PII(D2,5,8,12): Missing | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PII(D5,8,12,14): Positive | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PII(D5,8,12,14): Undetermined | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PII(D5,8,12,14): Negative | 100 | 100 | 100
  DEN-4, RNA - PII(D5,8,12,14): Missing | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PII(M7): Positive | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PII(M7): Undetermined | 0.0 | 0.0 | 0.0
  DEN-4, RNA - PII(M7): Negative | 100 | 100 | 100
  DEN-4, RNA - PII(M7): Missing | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | T-DEN F17 | T-DEN F19 | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 2/40 | 1/40
Other Adverse Events (participants affected / at risk) | 39/40 | 34/40 | 35/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DEN F17 (N=40) | T-DEN F19 (N=40) | Placebo Comparator (N=40)
Eptopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DEN F17 (N=40) | T-DEN F19 (N=40) | Placebo Comparator (N=40)
Pain (General disorders) | 19 (19) | 10 (10) | 10 (10) — Dose 1
Redness (Skin and subcutaneous tissue disorders) | 16 (16) | 15 (15) | 9 (9) — Dose 1
Swelling (General disorders) | 9 (9) | 6 (6) | 5 (5) — Dose 1
Abdonimal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3) — Dose 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 1 (1) — Dose 1
Fatigue (General disorders) | 25 (25) | 16 (16) | 14 (14) — Dose 1
Fever (General disorders) | 13 (13) | 10 (10) | 10 (10) — Dose 1
Headache (Nervous system disorders) | 22 (22) | 10 (10) | 11 (11) — Dose 1
Muscle aches (Musculoskeletal and connective tissue disorders) | 15 (15) | 9 (9) | 9 (9) — Dose 1
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 3 (3) — Dose 1
Pain behind eyes (Eye disorders) | 15 (15) | 7 (7) | 7 (7) — Dose 1
Photophobia (Eye disorders) | 3 (3) | 1 (1) | 1 (1) — Dose 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 4 (4) — Dose 1
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 2 (2) — Dose 1
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — Dose 1
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) — Dose 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) — Dose 2
Fatigue (General disorders) | 16 (16) | 6 (6) | 7 (7) — Dose 2
Fever (General disorders) | 9 (9) | 9 (9) | 6 (6) — Dose 2
Headache (Nervous system disorders) | 18 (18) | 4 (4) | 8 (8) — Dose 2
Muscle aches (Musculoskeletal and connective tissue disorders) | 12 (12) | 2 (2) | 4 (4) — Dose 2
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) — Dose 2
Pain behind eyes (Eye disorders) | 8 (8) | 1 (1) | 3 (3) — Dose 2
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 2 (2) — Dose 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 4 (4) — Dose 2
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) — Dose 2
Vomitng (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Dose 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Consitpation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (4) | 2 (2)
Pharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0) | 4 (4)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 7 (7) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Venipuncture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No